CLINICAL TRIAL: NCT00733135
Title: Determination of Safety and Effectiveness of the SilverHawk™ Peripheral Plaque Excision System for Calcium (SilverHawk LS-C) and the SpiderFX™ Embolic Protection Device for the Treatment of Calcified Peripheral Arterial Disease in the Superficial Femoral and/or the Popliteal Arteries (DEFINITIVE Ca++)
Brief Title: Study of the SilverHawk™ /TurboHawk™ Plaque Excision Systems Used With SpiderFX to Treat Calcified Peripheral Arterial Disease (DEFINITIVE Ca++)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FHT-P-07-003
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral vascular disease; atherectomy; atherosclerosis; calcified lesions
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atherectomy with embolic protection (Other): All subjects were treated with atherectomy (with SilverHawk or TurboHawk device) in conjunction with embolic protection (SpiderFX device).
  Interventions: Device: SilverHawk™ LS-C, TurboHawk™ LS-C, TurboHawk™ LX-C plaque excision systems and SpiderFX™ embolic protection device

INTERVENTIONS:
Device: SilverHawk™ LS-C, TurboHawk™ LS-C, TurboHawk™ LX-C plaque excision systems and SpiderFX™ embolic protection device — Catheter-based excision of moderate to severely calcified plaque located in the SFA and/or popliteal artery.

SUMMARY:
This is a multi-center, non-randomized, single arm study of the SilverHawk™ /TurboHawk™ plaque excision systems when used in conjunction with SpiderFX™ embolic protection device in treatment of moderate to severely calcified peripheral arterial disease in the superficial femoral and/or popliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent
* Willing to comply with follow-up evaluations at specified times
* Has leg pain due to peripheral arterial disease
* Disease located within the femoropopliteal artery
* Moderate to severe calcification

Exclusion Criteria:

* Previously implanted stent(s) or stent graft(s) in target leg
* Life expectancy less than 12 months
* Has any planned surgical or endovascular intervention of target vessel 30 days before or after index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clair, MD, Principal Investigator — The Cleveland Clinic; David Roberts, MD, Principal Investigator — Sutter Medical Center

REFERENCES:
- [Result] Roberts D, Niazi K, Miller W, Krishnan P, Gammon R, Schreiber T, Shammas NW, Clair D; DEFINITIVE Ca(+)(+) Investigators. Effective endovascular treatment of calcified femoropopliteal disease with directional atherectomy and distal embolic protection: final results of the DEFINITIVE Ca(+)(+) trial. Catheter Cardiovasc Interv. 2014 Aug 1;84(2):236-44. doi: 10.1002/ccd.25384. Epub 2014 Feb 5. PMID 24402764

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 133 subjects were enrolled in this study between October 30, 2008 and October 13, 2010. The type of location included hospitals with catheterization labs and/or vascular centers.
Groups:
- Study Cohort: All participants were treated with SilverHawk/TurboHawk atherectomy catheters, with the SpiderFX Embolic Protection Device placed distally.
Period: Overall Study
Arm/Group | Study Cohort
Started | 133
Completed | 131
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Study Cohort: All participants were treated with SilverHawk™ /TurboHawk™ plaque excision systems, with the SpiderFX™ embolic protection device placed distally.
Arm/Group | Study Cohort
Number analyzed (Participants) | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 95
Region of Enrollment [Number; unit: participants]
  United States | 133

OUTCOME MEASURES:

1. Primary Outcome: Successful Revascularization
Description: Less than or equal to 50% residual diameter stenosis following plaque excision remaining at the target lesion(s), as adjudicated by the angiographic core laboratory
Time Frame: at the end of the procedure
Population: Number of lesions assessed by the angiographic core lab
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Study Cohort
Number analyzed (Participants) | 133
Number analyzed (lesions) | 163
percentage of lesions | 92.0 [87.6 to 95.2]
Statistical Analysis 1: Comparison: Study Cohort; Test type: Superiority or Other; p < 0.05, GEE

2. Primary Outcome: Major Adverse Event Free Rate 30 Days
Description: MAE was defined as a serious adverse event that results in death, acute myocardial infarction, dissection (grade C or greater), clinical perforation, pseudo-aneurysm, thrombosis, distal embolism (clinically relevant), amputation, or clinically-driven target vessel revascularization (TVR), through 30 days post-procedure, as adjudicated by the Clinical Events Committee (CEC).
Time Frame: 30 Days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 131
percentage of participants | 93.1 [88.3 to 96.4]

3. Secondary Outcome: Technical Procedural Success
Description: Technical Procedural Success was defined as meeting all of the following requirements:
  * Less than or equal to 50% residual diameter stenosis at the target lesion(s), as adjudicated by the angiographic core laboratory
  * No procedure-related Major Adverse Events (MAE), as adjudicated by the Clinical Events Committee (CEC)
  * No device malfunction causing the procedure to be aborted
  * Successful delivery and placement of the SpiderFX™ embolic protection device
Time Frame: at the end of the procedure
Population: Total patient population minus one patient because there was no angiographic post-treatment core lab data available.
Measure: Number; unit: percentage of participants
Groups:
- Study Cohort: All participants were treated with SilverHawk/TurboHawk™ plaque excision systems with the SpiderFX™ embolic protection device placed distally.
Arm/Group | Study Cohort
Number analyzed (Participants) | 132
percentage of participants | 88.6

4. Secondary Outcome: Residual Diameter Stenosis
Description: This endpoint was met when there was less than 30% residual diameter stenosis following treatment with SilverHawk™ /TurboHawk™ plaque excision systems and any adjunctive therapy (if required), as adjudicated by the angiographic core laboratory.
Time Frame: at the end of the procedure
Population: 1 lesion not included because there is no angiographic core laboratory post-treatment data available
Measure: Number; unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Study Cohort
Number analyzed (Participants) | 133
Number analyzed (lesions) | 167
percentage of lesions | 64.1

5. Secondary Outcome: Presence of Debris in Deployed SpiderFx™ Embolic Protection Device
Description: Presence of debris in deployed SpiderFx™ embolic protection device
Time Frame: at the end of the procedure
Measure: Number; unit: percentage of deployed filters
Units Other Than Participants: deployed filters
Arm/Group | Study Cohort
Number analyzed (Participants) | 133
Number analyzed (deployed filters) | 138
percentage of deployed filters | 88.4

6. Secondary Outcome: Preservation of Run-off Distal to the Filter
Description: Preservation of run-off distal to SpiderFX™ distal embolic protection device was determined by angiography of run-off vessels at the end of the procedure, as adjudicated by the angiographic core laboratory.
Time Frame: at the end of the procedure
Population: 115/133 subjects had the required angiographic images to assess this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Study Cohort
Number analyzed (Participants) | 115
percentage of participants | 98.3

ADVERSE EVENTS:
Time Frame: Through 30 days post-procedure
Arm/Group | Study Cohort
Serious Adverse Events (participants affected / at risk) | 26/133
Other Adverse Events (participants affected / at risk) | 36/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Cohort (N=133)
Access Site AE (Vascular disorders) | 3 (3)
Amputation at or below metatarsal line (Vascular disorders) | 1 (1)
AV fistula, target vessel (Vascular disorders) | 1 (1)
Dissection, grade A or B; target vessel (Vascular disorders) | 4 (4)
Dissection, grade D or greater; target vessel (Vascular disorders) | 1 (1)
Distal embolism; plaque, thrombus (blood clot) or debris distal to the filter, clinically relevant (Vascular disorders) | 3 (3)
GI bleeding due to anticoagulation (Gastrointestinal disorders) | 1 (1)
Hypotension or hypertension (Vascular disorders) | 1 (1)
Myocardial infarction, acute (Vascular disorders) | 1 (1)
Renal insufficiency (Endocrine disorders) | 2 (2)
Pseudoaneurysm, non-target vessel (Vascular disorders) | 1 (1)
Target vessel revascularization; non-clinically driven (Vascular disorders) | 1 (1)
Thrombosis (acute and subacute); target vessel (Vascular disorders) | 1 (1)
Vessel clinical perforation, target vessel (Vascular disorders) | 3 (3)
Other, respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other (Surgical and medical procedures) | 7 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Cohort (N=133)
Access site adverse event (Vascular disorders) | 9 (10)
Dissection, grade A or B; target vessel (Vascular disorders) | 26 (26)
Other (Vascular disorders) | 24 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can not make any publication concerning the study without providing the sponsor 30 days to review it and provide comments. The Sponsor may require PI to delay publication until any factual errors are corrected. If the sponsor determines the proposed publication contains confidential information, or patentable subject matter that requires protection, the sponsor may require delay of the publication less than or equal to 90 days.